CLINICAL TRIAL: NCT05740202
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Efficacy of SHR-7367 in Subjects With Advanced Solid Tumors
Brief Title: A Trial of SHR-7367 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-7367-I-101
Record Dates: First submitted 2023-01-28; First posted 2023-02-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: The study was divided into three phases, the dose escalation phase and the dose extension phase and therapeutic effect extension of SHR-7367 in subjects with advanced malignant tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-7367 (Experimental)
  Interventions: Drug: SHR-7367

INTERVENTIONS:
Drug: SHR-7367 — The study was divided into three phases, the dose escalation phase and the dose extension phase and therapeutic effect extension of SHR-7367 in subjects with advanced malignant tumors.

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1 trial to evaluate the safety and tolerability of SHR-7367 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study;
2. Male or female aged ≥18 years and ≤75 years at the time of signing the ICF;
3. Histopathologically or cytologically documented advanced or metastatic malignancies;
4. At least 1 measurable lesion conforming to RECIST 1.1 criteria;
5. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
6. Female and male patients of reproductive potential must agree to use highly effective contraception.

Exclusion Criteria:

1. Any immunostimulants administered within 4 weeks;
2. Systemic anti-tumor therapy within 4 weeks;
3. Any investigational cancer therapy administered within 4 weeks;
4. Surgical procedures requiring general anesthesia within 4 weeks;
5. History of autoimmune diseases;
6. History of immunodeficiency;
7. Severe infections within 2 weeks prior to the first study treatment;
8. Clinically significant cardiovascular condition;
9. Prior malignancy (other than current malignant tumor) within 5 ears before the first dose of study treatment;
10. Known history of serious allergic reactions to the investigational product or its main ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Up to 3 weeks
  Number of participants with DLTs
Recommended phase II dose | first dose of study medication up to 21 days
  The Recommended phase II dose of SHR-7367 injection
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | Up to 12 months
  • Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Tumor response using RECIST 1.1 | From first dose to disease progression or death, whichever comes first, up to 12 months
peak time (Tmax) | Up to 12 months
peak concentration (Cmax) | Up to 12 months
area under curve from 0 to the last measurable concentration time point t (AUC0-t), | Up to 12 months
area under curve from 0 to infinity (AUC0-∞) | Up to 12 months
elimination half-life (t1/2) | Up to 12 months
clearance rate (CL) | Up to 12 months
steady-state apparent volume of distribution (Vss) | Up to 12 months
steady-state peak concentration (Cmax, ss) | Up to 12 months
steady-state valley concentration (Ctrough, ss) | Up to 12 months
accumulation ratio (Rac) | Up to 12 months
percentage of activated B lymphocyte subsets in peripheral blood | Up to 12 months
Immunogenicity index: drug-resistant antibody (ADA) | Up to 12 months
Efficacy endpoints: Objective response rate (ORR) | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided